CLINICAL TRIAL: NCT03611140
Title: Effect of a Dietary Portfolio (PD) (Nopal, Chia, Soy, Oat and Inulin) and Physical Activity on Gut Microbiota in Patients With Metabolic Syndrome
Brief Title: Effect of Functional Foods on Gut Microbiota in Metabolic Syndrome
Acronym: MetS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Nimbe Torres y Torres, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 793
Record Dates: First submitted 2018-07-25; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; gut microbiota; metabolic endotoxemia; functional foods
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: In the first stage, the participants with metabolic syndrome consumed a reduced-energy diet tailored to provide a 500 kcal/d deficit as recommended by NIH with respect to their habitual diet for 15 days. In the second stage, the participants continued to consume the reduced energy diet with the addition of a combination of functional foods (dietary portfolio; DP). The DP provided 200 kcal that were subtracted from the diet. The kcal, appearance, and flavor were similar in DP and P. The DP and P were given in a package in a dehydrated form ready to be dissolved in water. The DP was divided into two packages, the first package contained 30 g of DP o P given in the breakfast and dissolved in 250ml and the second package was given at the dinner time and contained 30 g of P and DP dissolved in 250 mL of water.
Who Masked: Participant, Investigator
Masking Description: PD and placebo interventions were packaged identically in appearance, both the researcher and the participant did not know what type of maneuver was assigned. The packages were distributed by a person outside the study who was the same person who performed the randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary portfolio (DP) (Experimental): The dietary portfolio was given daily at the breakfast and dinner for 2 months. The dietary intervention was a combination of functional foods (dehydrated nopal, chia seed, soy protein, oat, and inulin) that was provided in a dehydrated form in packages of 30 g dissolved in 250 ml water for breakfast and 30 g in 250ml water for dinner.
  Interventions: Dietary Supplement: DP
- placebo (P) (Placebo Comparator): The placebo (P) was given daily at the breakfast and dinner for 2 months. The placebo intervention consisted of a mixture of calcium caseinate, maltodextrins, sweetener and of artificial flavoring that was provided in a dehydrated form in packages of 30 g dissolved in 250 ml water for breakfast and 30 g in 250ml water for dinner.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DP — a package containing a mix of functional foods
  Arms: Dietary portfolio (DP)
Dietary Supplement: Placebo — a package containing maltodextrins and caseinate calcium to mimic the DP
  Arms: placebo (P)

SUMMARY:
Aim: To study the effect of a combination of functional foods on gut microbiota in subjects with metabolic syndrome. Subjects that met the metabolic syndrome criteria were enrolled in a double-blind, parallel-arm, placebo-control study. The subjects were randomized to receive a dietary portfolio (DP) or placebo (P) treatment for 2 mo. The primary endpoint was to study the effect of a DP on gut microbiota. Secondary endpoints were biochemical and anthropometric parameters, LPS, insulin, leptin, area under the curve for glucose and insulin.

DETAILED DESCRIPTION:
This study was a single-center, randomized, controlled, double-blind, parallel versus placebo that consisted of five visits. The first visit was a screening evaluation to determine whether subjects met the inclusion criteria. The selected subjects were invited to a second visit that consisted of a medical history, 2-h oral glucose tolerance test (OGTT), the collection of stool samples for DNA isolation and collection of 5 ml blood sample. The participants received during the first stage, a low saturated fat diet (LSFD) for 15 days. In the third visit and second stage of dietary treatment, subjects were randomized to receive the dietary portfolio (DP) or placebo (P) treatment + an LSFD accompanied of a reduced energy diet for 1 mo. In the fourth visit, with a 1 mo interval, dietary assessment and compliance to the DP or P were evaluated. During each follow-up visit, a 24-h dietary recall was collected, a physical activity questionnaire was filled out and anthropometric and clinical parameters were assessed. In the fifth visit, a 2 -h oral glucose tolerance test (OGTT) was performed, and a stool sample for DNA isolation and 5 ml blood were collected.

Dietary intervention in the first stage, the participants consumed a reduced-energy diet tailored to provide a 500-kcal/d deficit as recommended by NIH with respect to their habitual diet for 15 days. The diet plan consisted in 50-60% carbohydrates, 15% protein, 25-35% fat, <7% saturated fat, ≤ 200 mg, 20-35 g fiber, 2000 mg/d sodium based on total energy. In the second stage, the participants continued to consume the reduced energy diet with the addition of a combination of functional foods (DP). The DP provided 200 kcal that were subtracted from the diet. The DP consisted of a mixture of 14 g de dehydrated nopal, 4 g of chia, 25 g of soy protein, 14 g of oat, 4 g of inulin, 0.15 of flavoring. The placebo (P) consisted of 30 g of calcium caseinate, 30 g of maltodextrin and 0.2 g of flavoring. The kcal, appearance, and flavor were similar in DP and P. The DP and P were given in a package in the dehydrated form ready to be dissolved in water. The DP was divided into two packages, the first package contained 17.3 g of DP or P given in the breakfast and dissolved in 250 ml and the second package was given at the dinner time, and contained 34.7 g of P and DP dissolved in 300 ml of water.

Dietary compliance. Dietary compliance was assessed with a 24-h dietary recall and 3-d food record (food lo), during each visit that was analyzed by food processor nutrition analysis software. The compliance of the consumption of the DP or P was evaluated with the number of empty packages returned at the following visit. Physical activity was assessed using the International physical activity questionnaire (IPAQ)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for controls (healthy)
* Male or female
* Adults between 20 and 60 years old
* BMI ≥ 20 to ≤ 25 kg/m2
* Patients with no criteria positive metabolic syndrome
* Patients who knew how to read and write
* Signature of informed consent

Inclusion Criteria of cases

* Male or female
* Adults between 20 and 60 years old
* BMI ≥ 25to ≤ 50 kg/m2
* Patients with 3 positive criteria of the metabolic syndrome
* Glucose > 100 to < 126 mg / dl
* Triglycerides > 150 mg / dl
* HDL-cholesterol: men < 40mg / dl and women <50 mg / dl
* Waist circumference > 80cm in women and> 90 cm in men
* Blood pressure ≥ 130/85 mmHg (in two different days)
* Patients who knew how to read and write
* Signature of informed consent

Exclusion Criteria:

* - Patients with any type of diabetes.
* Diseases that produce secondary obesity or diabetes
* Cardiovascular event
* Weight loss > 3 kgs in the last 3 months after the evaluation of the criteria
* Catabolic diseases such as cancer and acquired immunodeficiency syndrome
* Gravity status
* Positive smoking
* Treatment with medications

  * Treatment with antihypertensive drugs
  * Treatment with hypoglycemic agents or insulin and antidiabetics.
  * Treatment with statins, fibrates or other drugs to control the dyslipidemia.
  * Use of steroid medications, chemotherapy, immunosuppressants or radiotherapy.
  * Anorexigens or accelerate weight loss.
  * Any drug or medication that activates intestinal motility
  * Laxatives or antispasmodics 4 weeks before the study
  * Treatment with antibiotics 2 months before the study
* Patients with a digestive functional disorder (constipation, diarrhea, dyspepsia, functional abdominal distension) (determined by questionnaire based on the classification of Rome II).
* Inflammatory bowel disease
* Irritable bowel syndrome or other chronic gastrointestinal diseases
* Major surgery
* Treatment with pro / pre / symbiotic
* High fiber foods consumption (more than 15 grams of fiber)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiota | change after 2.5 months of dietary intervention with respect to baseline
  Fecal samples were collected to isolate DNA and sequenced using the Illumina platform

SECONDARY OUTCOMES:
glucose | change after 2.5 months of dietary intervention with respect to baseline
  serum glucose (mg/dl)
insulin | change after 2.5 months of dietary intervention with respect to baseline
  serum insulin (µU/ml)
glycated hemoglobin | change after 2.5 months of dietary intervention with respect to baseline
  plasma glycated hemoglobin (HbA1c) (%)
triglycerides | change after 2.5 months of dietary intervention with respect to baseline
  serum triglycerides (mg/dl)
cholesterol | change after 2.5 months of dietary intervention with respect to baseline
  serum total cholesterol (mg/dl)
LDL cholesterol | change after 2.5 months of dietary intervention with respect to baseline
  serum LDL- cholesterol (mg/dl)
HDL cholesterol | change after 2.5 months of dietary intervention with respect to baseline
  serum HDL- cholesterol (mg/dl)
LPS | change after 2.5 months of dietary intervention with respect to baseline
  lipopolysaccharide (LPS) (ng/ml)
CRP | change after 2.5 months of dietary intervention with respect to baseline
  serum C reactive protein (CRP) (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Nimbe y Torres, PhD, Principal Investigator — Instituto Nacional de Ciencias Médicas y Nutrición
Locations (1):
- Nimbe Torres y Torres, Mexico City, Please Select An Option Below, Mexico

REFERENCES:
- [Background] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Result] Ando K, Fujita T. Metabolic syndrome and oxidative stress. Free Radic Biol Med. 2009 Aug 1;47(3):213-8. doi: 10.1016/j.freeradbiomed.2009.04.030. Epub 2009 May 3. PMID 19409982
- [Result] Hansel B, Kontush A, Bonnefont-Rousselot D, Bruckert E, Chapman MJ. Alterations in lipoprotein defense against oxidative stress in metabolic syndrome. Curr Atheroscler Rep. 2006 Nov;8(6):501-9. doi: 10.1007/s11883-006-0026-8. PMID 17045077
- [Result] Guevara-Cruz M, Tovar AR, Aguilar-Salinas CA, Medina-Vera I, Gil-Zenteno L, Hernandez-Viveros I, Lopez-Romero P, Ordaz-Nava G, Canizales-Quinteros S, Guillen Pineda LE, Torres N. A dietary pattern including nopal, chia seed, soy protein, and oat reduces serum triglycerides and glucose intolerance in patients with metabolic syndrome. J Nutr. 2012 Jan;142(1):64-9. doi: 10.3945/jn.111.147447. Epub 2011 Nov 16. PMID 22090467
- [Result] Lopez-Romero P, Pichardo-Ontiveros E, Avila-Nava A, Vazquez-Manjarrez N, Tovar AR, Pedraza-Chaverri J, Torres N. The effect of nopal (Opuntia ficus indica) on postprandial blood glucose, incretins, and antioxidant activity in Mexican patients with type 2 diabetes after consumption of two different composition breakfasts. J Acad Nutr Diet. 2014 Nov;114(11):1811-8. doi: 10.1016/j.jand.2014.06.352. Epub 2014 Aug 12. PMID 25132122
- [Result] Torres N, Guevara-Cruz M, Granados J, Vargas-Alarcon G, Gonzalez-Palacios B, Ramos-Barragan VE, Quiroz-Olguin G, Flores-Islas IM, Tovar AR. Reduction of serum lipids by soy protein and soluble fiber is not associated with the ABCG5/G8, apolipoprotein E, and apolipoprotein A1 polymorphisms in a group of hyperlipidemic Mexican subjects. Nutr Res. 2009 Oct;29(10):728-35. doi: 10.1016/j.nutres.2009.09.013. PMID 19917453
- [Result] Jenkins DJ, Josse AR, Wong JM, Nguyen TH, Kendall CW. The portfolio diet for cardiovascular risk reduction. Curr Atheroscler Rep. 2007 Dec;9(6):501-7. doi: 10.1007/s11883-007-0067-7. PMID 18377791
- [Result] Ascencio C, Torres N, Isoard-Acosta F, Gomez-Perez FJ, Hernandez-Pando R, Tovar AR. Soy protein affects serum insulin and hepatic SREBP-1 mRNA and reduces fatty liver in rats. J Nutr. 2004 Mar;134(3):522-9. doi: 10.1093/jn/134.3.522. PMID 14988441
- [Result] Sanchez-Tapia M, Aguilar-Lopez M, Perez-Cruz C, Pichardo-Ontiveros E, Wang M, Donovan SM, Tovar AR, Torres N. Nopal (Opuntia ficus indica) protects from metabolic endotoxemia by modifying gut microbiota in obese rats fed high fat/sucrose diet. Sci Rep. 2017 Jul 5;7(1):4716. doi: 10.1038/s41598-017-05096-4. PMID 28680065
- [Result] Roberfroid MB. Prebiotics and probiotics: are they functional foods? Am J Clin Nutr. 2000 Jun;71(6 Suppl):1682S-7S; discussion 1688S-90S. doi: 10.1093/ajcn/71.6.1682S. PMID 10837317
- [Result] Turnbaugh PJ, Ridaura VK, Faith JJ, Rey FE, Knight R, Gordon JI. The effect of diet on the human gut microbiome: a metagenomic analysis in humanized gnotobiotic mice. Sci Transl Med. 2009 Nov 11;1(6):6ra14. doi: 10.1126/scitranslmed.3000322. PMID 20368178
- [Derived] Guevara-Cruz M, Flores-Lopez AG, Aguilar-Lopez M, Sanchez-Tapia M, Medina-Vera I, Diaz D, Tovar AR, Torres N. Improvement of Lipoprotein Profile and Metabolic Endotoxemia by a Lifestyle Intervention That Modifies the Gut Microbiota in Subjects With Metabolic Syndrome. J Am Heart Assoc. 2019 Sep 3;8(17):e012401. doi: 10.1161/JAHA.119.012401. Epub 2019 Aug 27. PMID 31451009